CLINICAL TRIAL: NCT03019289
Title: A Phase I, Open-Label, Single-Dose, Adaptive (S)-(-)-[18F]Fluspidine and [18F]Fallypride Positron Emission Tomography Study to Evaluate Sigma-1 and Dopamine-2 Receptor Occupancy by Pridopidine in the Human Brain of Healthy Volunteers and in Patients With Huntington's Disease
Brief Title: A Study to Evaluate Sigma-1 and Dopamine-2 Receptor Occupancy by Pridopidine in the Human Brain of Healthy Volunteers and in Patients With Huntington's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prilenia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TV7820-IMG-10082; 2016-001757-41 (EudraCT Number)
Record Dates: First submitted 2017-01-03; First posted 2017-01-12 (Estimated); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Health Volunteers, Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — pridopidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- pridopidine (Experimental): Pridopidine (TV-7820) capsules
  Interventions: Drug: pridopidine (90 mg)

INTERVENTIONS:
Drug: pridopidine (90 mg) — single dose will be administered in Cohort 1. Other optional cohorts 2 and 3 may include single dose 0.5 mg, 1 mg, 2.5 mg, 5 mg, 10 mg, 22.5 mg, 45 mg, or 90 mg. The dose will be selected based on the results obtained from Cohorts 1 and 2.

SUMMARY:
The purpose of this study is to demonstrate engagement of pridopidine with S1R and D2R (optional) in the living human brain. No formal statistical analysis will be conducted

ELIGIBILITY:
Inclusion Criteria:

* In general, good physical health as determined by medical history and psychiatric history, suicidality assessment & physical examination
* Men who are potentially fertile (not surgically [eg, vasectomy] or congenitally sterile
* Patients with Huntington's disease (HD): diagnosis of HD and with an onset of HD after 18 years of age

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The subject has been previously exposed to ionizing radiation or radioactive substances as a result of clinical research or medical treatment in the past 10 years.
* The subject has a counterindication to having an MRI
* History of alcohol, narcotic, or any other substance dependence in the past 2 years
* Additional Exclusion criteria to patients with Huntington's disease:
* The patient has a severe motor impairment that might cause artifacts.
* Patients with a known history of Long QT Syndrome or a first degree relative with this condition.
* Treatment with any investigational product within 6 weeks of screening or patients planning to participate in another clinical study assessing any investigational product during the study.

  * Additional criteria apply, please contact the investigator for more information

Min Age: 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Pharmaceuticals USA
Locations (1):
- Teva Investigational Site 32648, Leipzig, Germany

REFERENCES:
- [Background] Grachev ID, Meyer PM, Becker GA, Bronzel M, Marsteller D, Pastino G, Voges O, Rabinovich L, Knebel H, Zientek F, Rullmann M, Sattler B, Patt M, Gerhards T, Strauss M, Kluge A, Brust P, Savola JM, Gordon MF, Geva M, Hesse S, Barthel H, Hayden MR, Sabri O. Sigma-1 and dopamine D2/D3 receptor occupancy of pridopidine in healthy volunteers and patients with Huntington disease: a [18F] fluspidine and [18F] fallypride PET study. Eur J Nucl Med Mol Imaging. 2021 Apr;48(4):1103-1115. doi: 10.1007/s00259-020-05030-3. Epub 2020 Sep 29. PMID 32995944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers (HV) and patients with Huntington Disease (HD) were enrolled. The first participant was enrolled on 22 March 2017; the last subject completed the study on 09 February 2018.
Pre-assignment Details: The screening period had a duration of up to 8 weeks. A total of 49 healthy subjects and 3 HD patients were screened; of these, 20 healthy subjects and 3 HD patients met the eligibility criteria and were enrolled in the study.
Groups:
- A: Cohort 1: P90 + (S)-(-)-FPD; HV: Healthy volunteers (HV) receiving a single dose of 90 mg pridopidine (P90) and radiolabeled PET tracer (S)-(-)-[18F]fluspidine ((S)-(-)-FPD) for neuroimaging in Part A of the study
- A: Cohort 2: P45 + (S)-(-)-FPD; HV: Healthy volunteers (HV) receiving a single dose of 45 mg pridopidine (P45) and radiolabeled PET tracer (S)-(-)-[18F]fluspidine ((S)-(-)-FPD) for neuroimaging in Part A of the study
- A: Cohort 2: P22.5 + (S)-(-)-FPD; HV: Healthy volunteers (HV) receiving a single dose of 22.5 mg pridopidine (P22.5) and radiolabeled PET tracer (S)-(-)-[18F]fluspidine ((S)-(-)-FPD) for neuroimaging in Part A of the study
- A: Cohort 3: P5 + (S)-(-)-FPD; HV: Healthy volunteers (HV) receiving a single dose of 5 mg pridopidine (P5) and radiolabeled PET tracer (S)-(-)-[18F]fluspidine ((S)-(-)-FPD) for neuroimaging in Part A of the study
- A: Cohort 7: P1 + (S)-(-)-FPD; HV: Healthy volunteers (HV) receiving a single dose of 1 mg pridopidine (P1) and radiolabeled PET tracer (S)-(-)-[18F]fluspidine ((S)-(-)-FPD) for neuroimaging in Part A of the study
- A: Cohort 7: P0.5 + (S)-(-)-FPD; HV: Healthy volunteers (HV) receiving a single dose of 0.5 mg pridopidine (P0.5) and radiolabeled PET tracer (S)-(-)-[18F]fluspidine ((S)-(-)-FPD) for neuroimaging in Part A of the study
- A: Cohort 6; P90 + (S)-(-)-FPD; HD: Patients with Huntington's Disease (HD) receiving a single dose of 90 mg pridopidine (P90) and radiolabeled PET tracer (S)-(-)-[18F]fluspidine ((S)-(-)-FPD) for neuroimaging in Part A of the study
- B: Cohort 4: P90 + Fallypride; HV: Healthy volunteers (HV) receiving a single dose of 90 mg pridopidine (P90) and radiolabeled PET tracer [18F]fallypride for neuroimaging in Part B of the study
- Cohort 0: (S)-(-)-FPD, HV: Healthy volunteers (HV) receiving a single dose of radiolabeled PET tracer (S)-(-)-[18F]fluspidine ((S)-(-)-FPD) for neuroimaging
Period: Overall Study
Arm/Group | A: Cohort 1: P90 + (S)-(-)-FPD; HV | A: Cohort 2: P45 + (S)-(-)-FPD; HV | A: Cohort 2: P22.5 + (S)-(-)-FPD; HV | A: Cohort 3: P5 + (S)-(-)-FPD; HV | A: Cohort 7: P1 + (S)-(-)-FPD; HV | A: Cohort 7: P0.5 + (S)-(-)-FPD; HV | A: Cohort 6; P90 + (S)-(-)-FPD; HD | B: Cohort 4: P90 + Fallypride; HV | Cohort 0: (S)-(-)-FPD, HV
Started | 5 | 1 | 3 | 2 | 1 | 1 | 3 | 4 | 3
Completed | 3 | 1 | 3 | 2 | 1 | 1 | 3 | 4 | 2
Not Completed | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects/patients enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Cohort 1: P90 + (S)-(-)-FPD; HV | A: Cohort 2: P45 + (S)-(-)-FPD; HV | A: Cohort 2: P22.5 + (S)-(-)-FPD; HV | A: Cohort 3: P5 + (S)-(-)-FPD; HV | A: Cohort 7: P1 + (S)-(-)-FPD; HV | A: Cohort 7: P0.5 + (S)-(-)-FPD; HV | A: Cohort 6; P90 + (S)-(-)-FPD; HD | B: Cohort 4: P90 + Fallypride; HV | Cohort 0: (S)-(-)-FPD, HV | Total
Number analyzed (Participants) | 5 | 1 | 3 | 2 | 1 | 1 | 3 | 4 | 3 | 23
Age, Continuous [Median (Full Range); unit: years] | 28.0 [27 to 30] | 26.0 [26 to 26] | 25.0 [25 to 28] | 27.5 [27 to 28] | 30 [30 to 30] | 25.0 [25 to 25] | 40.0 [32 to 58] | 28.0 [25 to 35] | 29.0 [25 to 30] | 28 [25 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 3 | 2 | 1 | 1 | 3 | 4 | 3 | 23
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 1 | 3 | 2 | 1 | 1 | 3 | 4 | 2 | 22
  Black/African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Germany | 5 | 1 | 3 | 2 | 1 | 1 | 3 | 4 | 3 | 23

OUTCOME MEASURES:

1. Primary Outcome: Sigma-1 Receptor Occupancy
Description: Receptor occupancy of pridopidine to Sigma-1 receptors (S1R) in the brain was assessed from Positron Emission Tomography (PET) imaging with (S)-(-)-[18F]fluspidine
Time Frame: 2 hours after oral administration of pridopidine
Population: Patients enrolled and receiving pridopidine. Patients from Cohort B (receiving fallypride only) and Cohort 0 (no pridopidine treatment) were not included in the analysis
Measure: Mean (Full Range); unit: percentage of receptor occupancy
Arm/Group | A: Cohort 1: P90 + (S)-(-)-FPD; HV | A: Cohort 2: P45 + (S)-(-)-FPD; HV | A: Cohort 2: P22.5 + (S)-(-)-FPD; HV | A: Cohort 3: P5 + (S)-(-)-FPD; HV | A: Cohort 7: P1 + (S)-(-)-FPD; HV | A: Cohort 7: P0.5 + (S)-(-)-FPD; HV | A: Cohort 6; P90 + (S)-(-)-FPD; HD
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 1 | 1 | 3
percentage of receptor occupancy | 91.21 [88.82 to 95.67] | 87.19 [87.19 to 87.19] | 86.67 [84.06 to 89.24] | 77.96 [76.75 to 79.16] | 41.77 [41.77 to 41.77] | 17.55 [17.55 to 17.55] | 87.37 [80.36 to 93.23]

2. Secondary Outcome: Maximum Plasma Concentration of Pridopidine
Description: Maximum plasma concentration of pridopidine based on noncompartmental analysis
Time Frame: PK sampling 1 h before pridopidine dosing, and 5, 15, 30, 45, 60 min, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 h after dosing.
Population: Patients enrolled who received pridopidine and had sufficient data to calculate at least 1 evaluable pharmacokinetic parameter for pridopidine.
Measure: Geometric Mean (Full Range); unit: ng/mL
Groups:
- B: Cohort 4: P90 + FPD; HV: Healthy volunteers (HV) receiving a single dose of 90 mg pridopidine (P90) and radiolabeled PET tracer [18F]fallypride for neuroimaging in Part B of the study
Arm/Group | A: Cohort 1: P90 + (S)-(-)-FPD; HV | A: Cohort 2: P45 + (S)-(-)-FPD; HV | A: Cohort 2: P22.5 + (S)-(-)-FPD; HV | A: Cohort 3: P5 + (S)-(-)-FPD; HV | A: Cohort 7: P1 + (S)-(-)-FPD; HV | A: Cohort 7: P0.5 + (S)-(-)-FPD; HV | A: Cohort 6; P90 + (S)-(-)-FPD; HD | B: Cohort 4: P90 + FPD; HV
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 1 | 1 | 3 | 4
ng/mL | 552 [496 to 614] | 307 [307 to 307] | 147 [117 to 184] | 25.9 [16.1 to 41.8] | 2.90 [2.90 to 2.90] | 1.33 [1.33 to 1.33] | 764 [666 to 877] | 452 [244 to 724]

3. Secondary Outcome: Time to Reach Maximum (Peak) Concentration (Tmax)
Description: Multiple PK samples over 24 hours will be calculated for pridopidine and its metabolite TV-45065 in plasma using non-compartmental methods, when possible.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | A: Cohort 1: P90 + (S)-(-)-FPD; HV | A: Cohort 2: P45 + (S)-(-)-FPD; HV | A: Cohort 2: P22.5 + (S)-(-)-FPD; HV | A: Cohort 3: P5 + (S)-(-)-FPD; HV | A: Cohort 7: P1 + (S)-(-)-FPD; HV | A: Cohort 7: P0.5 + (S)-(-)-FPD; HV | A: Cohort 6; P90 + (S)-(-)-FPD; HD | B: Cohort 4: P90 + Fallypride; HV
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 1 | 1 | 3 | 4
hours | 1.97 [1.50 to 3.00] | 1.98 [1.98 to 1.98] | 1.00 [0.75 to 1.50] | 1.00 [0.75 to 1.50] | 1.98 [1.98 to 1.98] | 1.97 [1.97 to 1.97] | 1.00 [0.50 to 1.62] | 2.26 [1.00 to 5.02]

4. Other Pre Specified Outcome: Dopamine-2 Receptor Occupancy
Description: RO of D2 (Dopamine-2) at 2 hours after oral administration of pridopidine (90 mg dose level) was investigated in 4 healthy volunteers using [18F]fallypride
Time Frame: 2 h after pridopidine dosing
Population: Patients enrolled and treated
Measure: Mean (Standard Deviation); unit: percent volume/volume
Arm/Group | B: Cohort 4: P90 + FPD; HV
Number analyzed (Participants) | 4
percent volume/volume | 3.34 (2.05)

ADVERSE EVENTS:
Time Frame: From signing of the informed consent through to 7 days after the last administration of study drug.
Arm/Group | A: Cohort 1: P90 + (S)-(-)-FPD; HV | A: Cohort 2: P45 + (S)-(-)-FPD; HV | A: Cohort 2: P22.5 + (S)-(-)-FPD; HV | A: Cohort 3: P5 + (S)-(-)-FPD; HV | A: Cohort 7: P1 + (S)-(-)-FPD; HV | A: Cohort 7: P0.5 + (S)-(-)-FPD; HV | A: Cohort 6; P90 + (S)-(-)-FPD; HD | B: Cohort 4: P90 + Fallypride; HV | Cohort 0: (S)-(-)-FPD, HV
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/1 | 0/3 | 0/2 | 0/1 | 0/1 | 0/3 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/1 | 0/3 | 0/2 | 0/1 | 0/1 | 0/3 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 2/5 | 1/1 | 1/3 | 0/2 | 0/1 | 0/1 | 1/3 | 1/4 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Cohort 1: P90 + (S)-(-)-FPD; HV (N=5) | A: Cohort 2: P45 + (S)-(-)-FPD; HV (N=1) | A: Cohort 2: P22.5 + (S)-(-)-FPD; HV (N=3) | A: Cohort 3: P5 + (S)-(-)-FPD; HV (N=2) | A: Cohort 7: P1 + (S)-(-)-FPD; HV (N=1) | A: Cohort 7: P0.5 + (S)-(-)-FPD; HV (N=1) | A: Cohort 6; P90 + (S)-(-)-FPD; HD (N=3) | B: Cohort 4: P90 + Fallypride; HV (N=4) | Cohort 0: (S)-(-)-FPD, HV (N=3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter site hematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site paraesthisia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sports injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data and results are owned by the sponsor. Results can be used by the institution for internal noncommercial research, education and patient care, and as required under applicable laws and regulations. Other uses require prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-05-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT03019289/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT03019289/SAP_001.pdf